CLINICAL TRIAL: NCT03629314
Title: Improving Surgical Patient Knowledge and Safe Use of Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jean Wong, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-5723
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Opioid Use
Keywords: Opioid

STUDY DESIGN:
Intervention Model Description: Educational-Interventional Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Pamphlet arm (Experimental): Educational Pamphlet will be provided to all participants to review, questionnaire will be provided to complete before and after review of the pamphlets
  Interventions: Other: Educational pamphlet arm

INTERVENTIONS:
Other: Educational pamphlet arm — Educational pamphlets will be provided to review and questionnaire will be provided to complete before and after review of the pamphlet

SUMMARY:
Opioids are commonly prescribed for surgical patients to treat moderate to severe pain after surgery. However, opioids can be associated with serious complications such as respiratory depression and death. Currently, it is not routine practice to educate surgical patients about the risks of opioids and how to safely use opioids after surgery. The investigators have developed an educational pamphlet specifically for surgical patients to educate them about the safe use of opioids. The objective of this pilot study is to determine the usability and readability of an educational pamphlet about the safe use, proper storage and disposal of opioids. The educational pamphlet will be modified based on the feedback from the pilot study and subsequently used for a randomized controlled trial.

DETAILED DESCRIPTION:
Twenty participants presenting to the preoperative clinic will be recruited for the pilot study. After informed consent is obtained, patients will be given an opioid knowledge questionnaire to complete before the education. They will then be given an educational pamphlet to review. After they have reviewed the educational pamphlet, they will complete the same opioid knowledge questionnaire. They will also complete a questionnaire evaluating the patient educational pamphlet. The pamphlet will be modified based on the feedback from the patients in the pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years adults
2. Proficient in English
3. scheduled for elective surgery

Exclusion Criteria:

1. Patients who are on opioids for chronic pain
2. Patients have taken opioids in the past 30 days
3. Patients who are unable to read and understand English -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Opioid Education Questionnaire | 10 - 15 minutes
  Total score 0-15 with higher scores representing more knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, MD, Principal Investigator — University Health Network/Toronto Western Hospital
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No